CLINICAL TRIAL: NCT03298256
Title: Three-dimensional Effects of Bracing in Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 15-493
Record Dates: First submitted 2017-09-25; First posted 2017-10-02 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: AIS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lenke type 1 AIS: Patients will be given a new prescription for a custom made Boston type thoracic-lumbo- sacral-orthosis (TLSO) braces. All patients will undergo low dose biplanar X-rays using the EOS ® machine system.
  Interventions: Radiation: EOS X-rays

INTERVENTIONS:
Radiation: EOS X-rays — Full length, orthogonal anteroposterior and lateral X-rays will be taken simultaneously in a standardised standing position, with arms folded anteriorly in 45 degrees . All radiographs will include C7 proximally and the femoral heads distally. 3D reconstruction of the spine can be performed. X-rays will be repeated after the brace is applied, and at intervals of no fewer than 6 months until the brace is weaned off, or if surgical intervention is required. Coronal, sagittal and axial parameters will be calculated from the reconstruction. 3D vertebral wedging will be calculated in the posterofrontal, sagittal and diagonal planes at the apex, 3 superior and 3 inferior vertebrae, as described by Scherrer et al. Changes in the pre- and post-bracing and follow-up parameters can be calculated.

SUMMARY:
This study intends to investigate the three dimensional (3D) effect of bracing on the adolescent idiopathic scoliosis (AIS). In particular, it will look at the relationship between frontal deformity correction and changes in the sagittal profile and apical vertebral rotation (AVR) during bracing. The investigators hypothesise that if the thoracic frontal deformity can be controlled with bracing, there will be spontaneous correction of the sagittal plane and rotation deformity through coupling.

DETAILED DESCRIPTION:
Scoliosis is a 3D deformity of the spine with curvatures occurring in three planes.

The efficacy of bracing in correcting the frontal deformity is now well-accepted after the Bracing in Adolescent Idiopathic Scoliosis Trial (BRAIST). Restoration of the sagittal alignment is one of the fundamental goals in scoliosis treatment. The investigators have previously demonstrated on fulcrum bending radiographs that there is coupling between the frontal deformity, thoracic kyphosis and apical vertebral derotation. The investigators' findings suggest that there may be natural coupling of the frontal and sagittal deformities towards "self-normalisation" during correction of the curves. The effect of bracing on the sagittal alignment and 3D deformity in scoliosis is currently not well-understood. If there is a tendency for the natural curve behaviour to return towards a more normal sagittal alignment, then bracing may exert a similar effect on the 3D profile. Understanding how the 3D deformity is affected by bracing allows further insight into curve progression and brace effectiveness.

Few studies in the literature have addressed the sagittal profile and 3D correction by bracing. Of those, the findings were based on vertebral reconstructions obtained from CT-scan, finite element analysis modelling, or studying the changes in the rib cage rotation. However, the investigators propose to measure the 3D profile using the modern EOS ® system, which allows biplanar radiography and 3D calculations and a more accurate measurement of vertebral wedging.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of Lenke type 1 AIS who fulfil the normal criteria for bracing

Exclusion Criteria:

* if the aetiology of the scoliosis is not idiopathic
* does not belong to Lenke type 1
* previous treatment with a brace
* severe presentation requiring surgical intervention
* unavailable for regular follow-up
* parents are unable to give informed consent

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted in the Department of Orthopaedics and Traumatology, The University of Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Compare change in three dimensional (3D) effect of bracing on the adolescent idiopathic scoliosis (AIS) using the EOS Imaging System | Follow-up to 3 years
  To compare change in full length, orthogonal anteroposterior and lateral X-rays in a standardised standing position after the brace is applied, and at intervals of no fewer than 6 months until the brace is weaned off, or if surgical intervention is required

SECONDARY OUTCOMES:
Measure health-related quality of life outcome by the 22-item Scoliosis Research Society questionnaire (SRS-22) of patients with adolescent idiopathic scoliosis (AIS) | Follow-up to 3 years
  To compare change in the health-related quality of life outcome of patients with adolescent idiopathic scoliosis (AIS) by the 22-item Scoliosis Research Society questionnaire (SRS-22), with the minimum score of 22 to the maximum score of 110. Higher score means better health outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kenny Kwan, BMBCh(Oxon), Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinstein SL, Dolan LA, Wright JG, Dobbs MB. Effects of bracing in adolescents with idiopathic scoliosis. N Engl J Med. 2013 Oct 17;369(16):1512-21. doi: 10.1056/NEJMoa1307337. Epub 2013 Sep 19. PMID 24047455
- [Background] Luk KD, Cheung WY, Wong Y, Cheung KM, Wong YW, Samartzis D. The predictive value of the fulcrum bending radiograph in spontaneous apical vertebral derotation in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2012 Jul 1;37(15):E922-6. doi: 10.1097/BRS.0b013e31824f108f. PMID 22744400
- [Background] Luk KD, Vidyadhara S, Lu DS, Wong YW, Cheung WY, Cheung KM. Coupling between sagittal and frontal plane deformity correction in idiopathic thoracic scoliosis and its relationship with postoperative sagittal alignment. Spine (Phila Pa 1976). 2010 May 15;35(11):1158-64. doi: 10.1097/BRS.0b013e3181bb49f3. PMID 20118836
- [Background] Parent S, Labelle H, Skalli W, de Guise J. Vertebral wedging characteristic changes in scoliotic spines. Spine (Phila Pa 1976). 2004 Oct 15;29(20):E455-62. doi: 10.1097/01.brs.0000142430.65463.3a. PMID 15480123
- [Background] Masharawi Y, Salame K, Mirovsky Y, Peleg S, Dar G, Steinberg N, Hershkovitz I. Vertebral body shape variation in the thoracic and lumbar spine: characterization of its asymmetry and wedging. Clin Anat. 2008 Jan;21(1):46-54. doi: 10.1002/ca.20532. PMID 17729333